CLINICAL TRIAL: NCT00292955
Title: An Exploratory Pharmacogenomic Study of Neoadjuvant Cetuximab Followed by Cisplatin, Radiotherapy, and Cetuximab in Women With Newly Diagnosed Locally Advanced or Metastatic Cervical Carcinoma
Brief Title: Cetuximab, Cisplatin, and Radiotherapy in Women With Locally Advanced Cervical Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: Bristol-Myers Squibb (Industry); Eli Lilly and Company (Industry); Washington University School of Medicine (Other)
Responsible Party: Linda R. Duska, M.D, University of Virginia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-HSR#13748; CA225243; HRPO #05-0702
Record Dates: First submitted 2006-02-14; First posted 2006-02-16 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Cancer of the Cervix
Keywords: Cervical Cancer, Cetuximab, Phase II Clinical Trials; Stage IB2-IVB Carcinoma of the Cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cetuximab

INTERVENTIONS:
Drug: Cetuximab — monotherapy (day 1), then weekly thereafter along with radiation. dose is at 200mg/m2.

SUMMARY:
The anti-tumor activity of cetuximab prior to chemoradiotherapy and the safety and tolerability of cetuximab with concurrent chemoradiation will be determined in women with locally advanced or metastatic cervical carcinoma.

DETAILED DESCRIPTION:
* Women with Federation of Gynecology and Obstetrics (FIGO) Clinical Stage IB2-IVB carcinoma of the cervix
* Baseline cervical biopsy, blood samples, and FDG-PET/computed tomography (CT) scan
* Cetuximab 400 mg/m2 on day 1 followed by cetuximab 250 mg/m2 on days 8 and 15
* Repeat cervical biopsy and FDG-PET/CT scan following cetuximab monotherapy
* Radiation and weekly cisplatin 40 mg/m2 and cetuximab 250 mg/2 for 6 weeks
* Cetuximab 250 mg/m2 weekly for 12 weeks
* Repeat cervical biopsy (if tumor present) and FDG-PET/CT scan after completion of therapy
* Follow for tumor recurrence and survival

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed a Washington University, Human Studies Committee (HSC) approved, informed consent.
2. Patients must have primary, histologically documented FIGO Clinical Stage IB2-IVB invasive carcinoma of the uterine cervix with measurable disease amendable to repeated biopsy.
3. Patients must have an ECOG performance status of 0, 1, or 2 at study entry.
4. Patients, 18 years and older, must either be not of child bearing potential or have a negative pregnancy test within 7 days of treatment. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal. Women should not breast feed while on this study.
5. Women must have a primary diagnosis of invasive carcinoma of the uterine cervix. Men are excluded from this study as a consequence of the diagnosis being investigated.
6. Patients must have had no previous treatment for invasive carcinoma of the uterine cervix.
7. Patients must be newly diagnosed with locally advanced or metastatic cervical carcinoma.
8. Bone marrow function: absolute neutrophil count (ANC) ≥ 1,500/mcl; platelets > 100,000/mcl.
9. Renal function: creatinine ≤ 2.0 mg/dl.
10. Hepatic function: bilirubin ≤ 1.5 times upper limit normal (ULN); SGOT ≤ 2.5 times upper limit normal (ULN).
11. Patients with ureteral obstruction must be treated with stent or nephrostomy tube placement.
12. Patients with neuropathy (sensory and motor) must be ≤ grade 1 defined by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 (June 10, 2003).

Exclusion Criteria:

1. Acute hepatitis or known HIV.
2. Active or uncontrolled infection.
3. Significant history of uncontrolled cardiac disease i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction.
4. Prior therapy which specifically and directly targets the EGFR pathway.
5. Prior severe infusion reaction to a monoclonal antibody.
6. Any concurrent chemotherapy not indicated in the study protocol or any other investigational agent(s).
7. A serious uncontrolled medical disorder that in the opinion of the Investigator would impair the ability of the subject to receive protocol therapy.
8. Unresolved ureteral obstruction.
9. Renal abnormalities, such as pelvic kidney, horseshoe kidney, or renal transplant, that would require modification of radiation fields.
10. Known or documented brain metastases.
11. Any concurrent malignancy other than non-melanoma skin cancer. (Patients with a previous malignancy but without evidence of disease for ≥ 5 years will be allowed to enter the trial).
12. Prior radiation therapy to the abdomen and/or pelvis
13. Incarceration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-02; Primary Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
To identify genes that may be identified as predictive of response to cetuximab | completion
To sequence the epidermal growth factor receptor (EGFR) to describe mutations in the receptor that may predict tumor response to cetuximab | completion
To evaluate the validity of fluorodeoxyglucose (FDG) uptake, as determined by positron emission tomography (PET) imaging, as a surrogate marker for response to cetuximab | completion

SECONDARY OUTCOMES:
To determine the safety and tolerability of cetuximab with concurrent chemoradiation in women with locally advanced cervical carcinoma | weekly
To determine the progression-free and overall survival in women with locally advanced or metastatic cervical carcinoma treated with concurrent chemoradiation and cetuximab | every three months

CONTACTS AND LOCATIONS:
Overall Officials: Linda R. Duska, M.D., Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - Washinton University School of Medicine, St Louis, Missouri
  - University of Virginia Cancer Center, Charlottesville, Virginia

REFERENCES:
- [Derived] Fracasso PM, Duska LR, Thaker PH, Gao F, Zoberi I, Dehdashti F, Siegel BA, Uliel L, Menias CO, Rehm PK, Goodner SA, Creekmore AN, Lothamer HL, Rader JS. An Exploratory Study of Neoadjuvant Cetuximab Followed by Cetuximab and Chemoradiotherapy in Women With Newly Diagnosed Locally Advanced Cervical Cancer. Am J Clin Oncol. 2022 Jul 1;45(7):286-293. doi: 10.1097/COC.0000000000000926. Epub 2022 Jun 7. PMID 35696702